CLINICAL TRIAL: NCT02168270
Title: A Phase I Study of Metronomic Temozolomide and Intravenous Ascorbic Acid for Patients With Recurrent High Grade Glioma
Brief Title: Temozolomide and Ascorbic Acid in Treating Patients With Recurrent High-Grade Glioma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: University of Nebraska (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0735-13-FB; NCI-2014-01061 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); P30CA036727 (NIH)
Record Dates: First submitted 2014-05-29; First posted 2014-06-20 (Estimated); Results first posted 2018-02-23 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Anaplastic Astrocytoma; Anaplastic Oligodendroglioma; Anaplastic Oligoastrocytoma; Glioblastoma; Gliosarcoma
MeSH Terms: conditions — Astrocytoma; Oligodendroglioma; Glioblastoma; Gliosarcoma | interventions — Ascorbic Acid; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment (ascorbic acid, temozolomide) (Experimental): Patients receive ascorbic acid IV over 90-120 minutes three times per week and temozolomide orally days 1-28. Treatment repeats every 4 weeks for up to 12 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Dietary Supplement: ascorbic acid; Drug: temozolomide; Other: quality-of-life assessment; Other: laboratory biomarker analysis

INTERVENTIONS:
Dietary Supplement: ascorbic acid — Given IV
  Other Names: C-Long; Ce-Vi-Sol; Cecon; Cenolate; Cetane
Drug: temozolomide — Given PO
  Other Names: SCH 52365; Temodal; Temodar; TMZ
Other: quality-of-life assessment — Ancillary studies
  Other Names: quality of life assessment
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase I trial studies the side effects and best dose of ascorbic acid when given together with temozolomide in treating patients with high-grade glioma that has come back. Drugs used in chemotherapy, such as temozolomide, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Ascorbic acid contains ingredients that may prevent or slow the growth of high-grade gliomas. Giving temozolomide with ascorbic acid may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the toxicities and determine the recommended dose of intravenous ascorbic acid given three times weekly in combination with temozolomide in patients with recurrent high grade glioma.

SECONDARY OBJECTIVES:

I. To evaluate changes in the levels of serum ascorbic acid using high-performance liquid chromatography (HPLC) with coulometric electrochemical detection) during therapy with ascorbic acid and temozolomide.

II. Radiographic assessment of disease status after 2 cycles of therapy with ascorbic acid and temozolomide.

III. To evaluate progression-free and overall survival of patients with recurrent high grade glioma treated with therapy with ascorbic acid and temozolomide.

IV. To descriptively examine quality of life (QOL) using European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaires (QLQ)-C30 during treatment.

OUTLINE: This is a dose-escalation study of ascorbic acid.

Patients receive ascorbic acid intravenously (IV) over 90-120 minutes three times per week and temozolomide orally days 1-28. Treatment repeats every 4 weeks for up to 12 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days, every 2 months for 1 year and then periodically thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have pathologically proven diagnosis of high grade glioma
* Patients must have received prior radiation therapy and standard temozolomide
* Patients must be three or more months from the end of chemoradiotherapy or have biopsy or imaging consistent with disease progression
* Patients must have recovered from toxicity of prior therapy
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2 or better
* Absolute neutrophil count (ANC) count >= 1,500/mm^3
* Hemoglobin >= 8 g/dL
* Platelet count >= 100,000/mm^3
* Serum creatinine that is at or below 2.0 mg/dL
* Serum aspartate aminotransferase (AST) and alanine aminotransferase (ALT) less than 1.5 times the upper limits of normal; note: if hepatic function is abnormal, the decision to initiate temozolomide treatment should carefully consider the benefits and risks for the individual patient
* Serum alkaline phosphatase less than 2.5 times the upper limits of normal; note: if hepatic function is abnormal, the decision to initiate temozolomide treatment should carefully consider the benefits and risks for the individual patient
* The patient must be aware of the neoplastic nature of his/her disease and willingly provide written, informed consent after being informed of the procedure to be followed, the experimental nature of the therapy, alternatives, potential benefits, side-effects, risks, and discomforts
* Women of reproductive potential must be non-pregnant and non-nursing and must agree to employ an effective barrier method of birth control throughout the study and for up to 6 months following treatment
* Women of child-bearing potential must have a negative pregnancy test within 7 days of initiating study; (no childbearing potential is defined as age 55 years or older and no menses for two years or any age with surgical removal of the uterus and/or both ovaries)

Exclusion Criteria:

* History of uncontrollable allergic reactions to temozolomide or ascorbic acid or to antiemetics appropriate for administration in conjunction with protocol-directed chemotherapy
* Known human immunodeficiency virus (HIV)-positivity AND actively being treated with highly active anti-retroviral therapy (HAART)
* History of glucose-6-phosphate dehydrogenase deficiency
* History of oxalate nephrolithiasis or urine oxalate > 60 mg/dL
* Anuria, dehydration, severe pulmonary congestion or pulmonary edema or fixed low cardiac input since all are conditions for which osmotic diuresis are contraindicated and ascorbic acid has high osmolarity
* Any other clinically significant medical disease or condition laboratory abnormality or psychiatric illness that, in the Investigator's opinion, may interfere with protocol adherence or a subject's ability to give informed consent
* Patients who are on the following drugs and cannot have a drug substitution: flecainide, methadone, amphetamines, quinidine, and chlorpropamide; note: high dose ascorbic acid may affect urine acidification and, as a result, may affect clearance rates of these drugs
* Simultaneous participation in other therapeutic clinical trials will not be allowed
* Inability to co-operate with the requirements of the protocol
* Pregnant and nursing women are excluded from this study

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2014-06-16 (Actual); Primary Completion 2015-08-20 (Actual); Study Completion 2015-08-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Shonka, MD, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Ascorbic Acid, Temozolomide)
Started | 4
Completed | 0
Not Completed | 4
Not completed — Lack of Efficacy | 4

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Ascorbic Acid, Temozolomide)
Number analyzed (Participants) | 4
Age, Continuous [Mean (Full Range); unit: years] | 42 [30 to 64]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose of Ascorbic Acid in Combination With Temozolomide
Description: Maximum tolerated dose of ascorbic acid in combination with temozolomide, defined as the highest dose tested which results in dose limiting toxicity (DLT) in no more than one of six evaluable patients. Graded by the National Cancer Institute (NCI) Common Toxicity Criteria for Adverse Events version 4.0. DLT incidence will be described by dose level.
Time Frame: 56 days
Population: This study was terminated as subjects had disease progression so no subjects were evaluable.
Arm/Group | Treatment (Ascorbic Acid, Temozolomide)
Number analyzed (Participants) | 0

2. Primary Outcome: Incidence Rates of Adverse Events, Graded According to the NCI Common Toxicity Criteria for Adverse Events Version 4.0
Description: The incidence rates of adverse events will be described by dose level. The frequency of occurrence of overall toxicity, categorized by toxicity grades, will be described.
Time Frame: Up to 30 days after last administration of study medication
Population: This study was terminated after only 4 patients enrolled. Incidence rates of adverse event could not be describe by dose level.
Arm/Group | Treatment (Ascorbic Acid, Temozolomide)
Number analyzed (Participants) | 0

3. Secondary Outcome: Changes in Serum Levels of Ascorbic Acid Using High-performance Liquid Chromatography (HPLC) With Coulometric Electrochemical Detection)
Description: Correlation of intracellular glutathione (in peripheral blood mononuclear cells) with ascorbic acid levels during therapy with ascorbic acid and temozolomide will be summarized using descriptive statistics to summarize changes over time.
Time Frame: Baseline to up to 52 weeks
Population: No patients were analyzed as all experienced progressive disease after 2 cycles of treatment.
Arm/Group | Treatment (Ascorbic Acid, Temozolomide)
Number analyzed (Participants) | 0

4. Secondary Outcome: Using Radiologic Measurements for Tumor Response
Description: The measurement of effect will be based on the Macdonald criteria
Time Frame: Up to 52 weeks
Population: This outcome measure was not analyzed as all patients had progressive disease by 2 cycles of treatment.
Arm/Group | Treatment (Ascorbic Acid, Temozolomide)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Up to 52 weeks
Arm/Group | Treatment (Ascorbic Acid, Temozolomide)
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 2/4
Other Adverse Events (participants affected / at risk) | 1/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Ascorbic Acid, Temozolomide) (N=4)
Headache (General disorders) | 1 (3)
Vomiting (Gastrointestinal disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (2)
Seizure (Nervous system disorders) | 1 (2)
Pain, Hip, back (Musculoskeletal and connective tissue disorders) | 1 (1)
Weakness (General disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Ascorbic Acid, Temozolomide) (N=4)
Lymphopenia (Blood and lymphatic system disorders) | 1 (2) — low lymphocyte count
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No